CLINICAL TRIAL: NCT04282434
Title: CLinical Epigenetic-sensitive trajectOries Underlying Pulmonary Arterial Hypertension and neTwoRk Analysis (CLEOPAHTRA)
Brief Title: DNA Methylation Dynamics Underlying Arterial Remodeling in PAH Patients: CLEOPAHTRA Clinical Trial
Acronym: CLEOPAHTRA
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator Giuditta Benincasa, University of Campania Luigi Vanvitelli
Other Study IDs: CLEOPAHTRA; PRIN2017F8ZB89 (Other Grant/Funding Number: Italian Ministry of University and Research (MIUR))
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Arterial Remodeling
Keywords: Adaptive immunity; DNA methylome; RNA-sequencing; Network analysis
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Vascular Remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Circulating T cells Lung tissue biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify epigenetic-sensitive modifications and novel biomarkers linked to pathogenesis of pulmonary arterial hypertension (PAH), we will perform the first study analyzing differentially-methylated regions (DMRs) in circulating T cells (CD04+ and CD08+) isolated from peripheral blood of patients undergoing right heart catheterization. Moreover, we will perform RNA deep sequencing on lung tissue biopsies to validate if DNA methylation signatures in circulating T cells could reflect perturbations of gene expression in lung tissues.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is characterized by remodeling of pulmonary arteries caused by an inbalance of proliferation/apoptosis rate within the vascular wall. This pathological phenotype seems to be triggered by different environmental stress and injury events such as increased inflammation, DNA damage, and epigenetic deregulation. Many immune cells are increased in PAH, such as T and B lymphocytes. Remarkably, T cells are essential players of adaptive immunity and may be relevant initiators ("initial hit") of vascular remodelling. We will perform the first multi-omics study to: 1) investigate DNA methylome of circulating T cells isolated from peripheral blood of PAH patients, 2) detect transcriptomic profiles of lung tissues, 3) to assess if DNA methylation of distinct genomic regions in circulating T cells could reflect modifications of lung gene expression programs.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with World Health Organization (WHO) Group I PAH.
* ≥ 18 years
* Documentation of the following hemodynamic parameters by right heart catheterization, performed at time of study enrolment:
* Mean pulmonary arterial pressure (mPAP) > 25 mmHg at rest or mPAP > 30 mm Hg with exercise.
* Pulmonary arterial wedge pressure (PAWP) ≤ 15 mm Hg.
* Pulmonary vascular resistance (PVR) ≥ 240 dynes.sec.cm-5 (e.g., ≥ 3.0 Wood units)

Exclusion Criteria:

* Patients who meet the criteria for inclusion into WHO Groups II, III, IV or V.
* Do not meet the required hemodynamic criteria for entry into the study.
* Patients with known history of cancer, malignancy disorders, active infections, and chronic or immune-mediated diseases.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 PAH patients (familial and idiopathic) vs 30 sex and age-matched subjects.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Identification of differentially methylated regions in CD04 and CD08 T cells | 3 Months
  Reduced Representation Bisulfite Sequencing
Identification of differentially expressed genes in lung tissue biopsies | 5 Months
  Chip Microarray
Bioinformatic analysis | 8 Months

CONTACTS AND LOCATIONS:
Overall Officials: Giuditta Benincasa, BiolD, MSc, Principal Investigator — University of Campania "L. Vanvitelli"
Locations (1):
- Monaldi Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Napoli C, Benincasa G, Loscalzo J. Epigenetic Inheritance Underlying Pulmonary Arterial Hypertension. Arterioscler Thromb Vasc Biol. 2019 Apr;39(4):653-664. doi: 10.1161/ATVBAHA.118.312262. PMID 30727752